CLINICAL TRIAL: NCT03964701
Title: Identification of Early Biomarkers of Peritoneal Membrane Dysfunction in Children on Peritoneal Dialysis Using Metabolomics Analysis
Brief Title: Peritoneal Membrane Dysfunction in Peritoneal Dialysis Using Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baxter (Hellas) Ltd (Industry)
Responsible Party: Principal Investigator, Nikoleta Printza, Associate Prof in Paediatric Nephrology, Aristotle University Of Thessaloniki
Other Study IDs: 98550
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: End Stage Renal Disease; Dialysis
Keywords: children; renal failure; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peritoneal dialysis PD effluent, blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no interventional study

SUMMARY:
Ability and sensitivity of metabolomics analysis to highlight biomarkers or a score of biomarkers that will be able to identify those pediatric patients on peritoneal dialysis at high risk for possible peritoneal dialysis complications and mainly encapsulating peritoneal sclerosis

DETAILED DESCRIPTION:
Ability and sensitivity of metabolomics analysis to highlight biomarkers or a score of biomarkers that will be able to identify those pediatric patients on peritoneal dialysis at high risk for possible peritoneal dialysis complications and mainly encapsulating peritoneal sclerosis. Identification of peritoneal membrane functional status changes over time, at the same patient (cohort study), by metabolomics, aiming in personalized medicine best practice.

Identification of peritoneal membrane functional status changes over time in immature infants' peritoneal membrane.

Identification of early and accurate markers of peritoneal membrane dysfunction when membrane status is possibly reversible that could predict peritoneal patients at risk for future loss of ultrafiltration and dialysis adequacy of small molecules examined today be PET, KT/V and Cr/Cl (when membrane status is not reversible).

Improve PD survival in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adolescent patients on peritoneal dialysis
* Aged:1month -20 years

Exclusion Criteria:

-Abdominal surgery

Ages: 30 Days to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Infants, children and adolescent patients on chronic peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-04-22 (Estimated); Study Completion 2020-04-22 (Estimated)

PRIMARY OUTCOMES:
Change of Peritoneal Equilibration test profile | 1 year
  Peritoneal Equilibration test

SECONDARY OUTCOMES:
Loss of dialysis adequency | 1 year
  KT/V
Elevated creatinine | 1 year
  Creatinine Clearence

CONTACTS AND LOCATIONS:
Overall Officials: Nikoleta Printza, Principal Investigator — Aristotle University
Locations (1):
- 1st ACADEMIC PEDIATRIC DEPARTMENT, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided